CLINICAL TRIAL: NCT06259591
Title: A Randomized, Controlled Trial to Evaluate if Pedometer-Guided Coaching Can Promote Postoperative Ambulation After Abdominopelvic Surgeries
Brief Title: Pedometer Coaching to Promote Postoperative Ambulation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Sergio D. Bergese, Director of Outcomes and Clinical Research in Perioperative Medicine, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB2022-00574
Record Dates: First submitted 2024-01-11; First posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Postoperative Outcomes
Keywords: Wearable Electronic Devices; Ambulation

STUDY DESIGN:
Masking Description: Pedometer data collection and coaching text administration will be done by an unmasked team member.
  30-day interview will be done by a masked team member.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pedometer follow-up and coaching (Experimental): Pedometer follow-up plus text message coaching Monday/ Wednesday/ Friday
  Interventions: Behavioral: Pedometer follow-up; Behavioral: Ambulation coaching
- Pedometer follow up (Active Comparator): Pedometer follow-up from day 8- 30 after surgery
  Interventions: Behavioral: Pedometer follow-up

INTERVENTIONS:
Behavioral: Pedometer follow-up — The daily step count will be obtained from the patients using a pedometer app (OutWalk) from day 8 to day 30 after surgery.
Behavioral: Ambulation coaching — Patients will receive coaching text messages every Monday, Wednesday and Friday between day 8 and day 30 after surgery, based on a pre-fixed template.
  Arms: Pedometer follow-up and coaching

SUMMARY:
The goal of this randomized controlled trial is to evaluate whether remote pedometer follow-up and virtual coaching can improve ambulation after major abdominopelvic surgery, and how this affects key postoperative outcomes.

The main questions it aims to answer are:

* Does pedometer-guided ambulation coaching increases ambulation after surgery?
* Does pedometer-guided coaching improve satisfaction, quality of recovery, while reducing postoperative complications?

Participants will be asked to install a pedometer app for the purpose of data sharing. Study personnel will compare pedometer follow-up plus text message coaching (intervention) with pedometer follow-up only (control) to investigate whether coaching improves adherence to the postoperative ambulation recommendation, and whether this leads to improvement of the secondary outcomes.

DETAILED DESCRIPTION:
Ambulation is not only a key component for improved postoperative recovery, studies have also found associations between the degree of ambulation in the early postoperative period and postoperative morbidity. Additionally, A preoperative sedentary lifestyle has been associated with a higher incidence of complications and readmissions after surgery . Our team conducted a systematic review, which found that perioperative pedometer readings were captured in 64-94% of the patients, and pedometer data were linked to a number of important perioperative outcomes including; complications; length of stay; and unplanned readmission. Several studies have demonstrated that inpatient pedometer-guided exercise programs could improve postoperative ambulation. However, this is limited by the length of hospital stay. In this study, the aim is to investigate the efficacy of pedometer-based coaching for post-discharge ambulation.

This is a randomized controlled trial with a 1:1 allocation ratio. Participants will be randomly allocated to either pedometer follow-up (control) or pedometer follow-up with 3 times per week ambulation coaching through texts (intervention). Participants will be screened and consented before surgery. All recruited subjects will have a pedometer app installed on their phone during the preoperative clinic visit, during which the purpose of the app and potential risks will be explained.

After surgery and confirmation of the postoperative criteria, participants will enter the study and undergo randomization through a automated system.

Postoperatively , participants in the control arm will have pedometer data collected over postoperative days 8-30. The participants in the interventional arm will also have the pedometer data collected, while additionally being provided feedback in the form of text message every Monday, Wednesday and Friday.

Pedometer data:

The pedometer app utilized for this study is called "Outwalk" and it is designed by a third party. The study team has a research account on the pedometer app. During the screening visit, after downloading the app and creating the deidentified study subject account, the subject enables their data to be shared with the research account. This provides automatic access to the step count data. The study team will have access to subject data and the unblinded team member will check the steps count.

The following details will be collected from the medical record and/or directly from the participants: Age, Gender , Race and Ethnicity, Planned surgery, American Society of Anesthesiologists (ASA) classification, Insurance status, BMI, Charlson comorbidity score, smoking status (never, former, current), alcohol status (never, social, regular), substance use disorder (yes or no), reports of postoperative delirium, unplanned admissions to emergency room or unplanned hospital visits after surgery,

The following are collected from the participants: Postoperative recovery satisfaction (1-10), Sleep quality (1-10), pre and postoperative Duke Activity Status Index (0-58.2), technical issues with pedometer or app use (no, or yes with explanation), Quality of Recovery 15 score (0-150)

Sample size:

Based on prior findings from prior studies, this study is expected to enroll 120 subjects (60 subjects per arm), accounting for loss to follow-up or restrictions of primary outcome. In an inpatient exercising program for patients undergoing laparoscopic surgery, the intervention increased step goal adherence from 7% to 27% with a sample size of 58 subjects per arm, Using 1:1 allocation with p<0.05 and power of 80%. In another study of open gynecology procedures; results showed the proportion of patients achieving activity goal (return to preoperative baseline) was 71% with pedometer-- based exercise intervention vs 41% control, with a sample size of 42 subjects per arm.

Participants who have missing data on more than 30% of the days will be removed from the study, their data will not be analyzed. Participants who have zero steps recorded for more than 30% of the days will also be treated as out-of-range results and will not be included in the primary analysis.

The investigation team plan to evaluate the distribution of the baseline characteristics between the two arms. Additional statistical analyses will be undertaken if there is significant baseline characteristics imbalance. Participants who have missing baseline data will be included in the primary and secondary analyses. The plan is to conduct a separate sensitivity analysis with these participants excluded. Participants with missing day 30 data will be included in the primary analyses. For such participants , any usable day-30 data will be included in the secondary analyses.

The primary analysis will compare the compliance with the ambulation goal between the coaching arm and the pedometer only arm. Compliance is defined as achieving at least 90% of the recommended ambulation goal (>2,250 steps per day), this is to accommodate for daily variation in activities, as well as to accommodate for missed step recording.

For the evaluation of secondary outcomes, the day 30 outcomes between the coaching arm and the pedometer follow-up arm will be compared. Additionally, the following exploratory analyses are planned:

1. Day-30 outcomes in participants who reached the ambulation goal compared to those who did not, including participants in both arms
2. Comparing the changes in daily step count across time from day 8 to day 30
3. Sensitivity analysis of primary outcome, where participants with out-of-range results will be included.
4. Sensitivity analysis of primary outcome, where participants with missing baseline data will be excluded.

Participants who have missing baseline data will be included in the primary and secondary analyses. A separate sensitivity analysis will be conducted with these patients excluded.

Participants with missing day 30 data will be included in the primary analyses. For such participants, any usable day-30 data will be included in the secondary analyses.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects ≥18 years at screening
* Subjects undergoing major abdominopelvic surgery under general anesthesia, expected to last more than 3 hours from induction of anesthesia to anesthesia stop time.
* Able to understand the study procedures and voluntarily provide study informed consent
* Agree to be followed up for the duration of the study period
* Has access to a smart phone with app compatibility
* Planned inpatient stay for 1 night or more

Exclusion Criteria:

* Subjects undergoing liver surgery or upper gastrointestinal surgery
* Refusal to install the app/ deleted app before end of the monitor period
* Subjects who are unable to walk at baseline
* Medical contraindications for unrestricted ambulation
* Patients with spinal or lower limb pathology, chronic or poorly controlled pain potentially preventing full postoperative ambulation
* Neurological impairment precluding unrestricted ambulation Cognitive impairment precluding consent or follow up study activities
* BMI >40
* Patients who require any mobility aid at baseline
* Subjects discharged to a rehab facility or never discharged from the hospital alive
* Hospital length of stay > 1 week
* Patient not cleared by physical therapy for unrestricted ambulation on discharge

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-01-31 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Adherence to ambulation goal | Postoperative day 8 to day 30
  Proportion of days on which patient met the ambulation goal

SECONDARY OUTCOMES:
30-day Duke Activity Status Index (DASI) score | Postoperative day 8 to day 30
  DASI score obtained through patient interview. This is a score which can range from 0 to 58.2. Higher score denotes better self-reported functional capacity.
30-day Quality of Recovery -15 (QoR-15) score | Postoperative day 8 to day 30
  QoR-15 score obtained through patient interview. This is a score which can range from 0-150. Higher score denotes better self-reported recovery after surgery.
Unplanned hospital visits | Postoperative day 8 to day 30
  Emergency room or hospital visits which are not part of the planned postoperative follow up visits, obtained through medical record review and patient interview
Sleep | Postoperative day 8 to day 30
  Quality of sleep. This is reported using a self-reported numerical rating scale which ranges from 0 to 10. Higher score denotes better sleep quality.
Patient satisfaction | Postoperative day 8 to day 30
  Patient satisfaction with the postoperative recovery. This is reported using a self-reported numerical rating scale which ranges from 0 to 10. Higher score denotes better satisfaction.
Postoperative delirium | Day of surgery to day of discharge (up to 7 days after surgery)
  Report of postoperative delirium during the hospital stay
Technical issue with the app or the follow up | Postoperative day 8 to day 30
  Patient reported issue with the pedometer app usage or the follow up process, obtained through patient interview

CONTACTS AND LOCATIONS:
Overall Officials: Sergio D Bergese, MD, FASA, Principal Investigator — Stony Brook Medicine
Locations (1):
- Stony Brook University Hospital, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hedrick TL, Hassinger TE, Myers E, Krebs ED, Chu D, Charles AN, Hoang SC, Friel CM, Thiele RH. Wearable Technology in the Perioperative Period: Predicting Risk of Postoperative Complications in Patients Undergoing Elective Colorectal Surgery. Dis Colon Rectum. 2020 Apr;63(4):538-544. doi: 10.1097/DCR.0000000000001580. PMID 32015289
- [Background] Nakajima H, Yokoyama Y, Inoue T, Nagaya M, Mizuno Y, Kayamoto A, Nishida Y, Nagino M. How Many Steps Per Day are Necessary to Prevent Postoperative Complications Following Hepato-Pancreato-Biliary Surgeries for Malignancy? Ann Surg Oncol. 2020 May;27(5):1387-1397. doi: 10.1245/s10434-020-08218-x. Epub 2020 Jan 23. PMID 31974713
- [Background] Bille A, Buxton J, Viviano A, Gammon D, Veres L, Routledge T, Harrison-Phipps K, Dixon A, Minetto MA. Preoperative Physical Activity Predicts Surgical Outcomes Following Lung Cancer Resection. Integr Cancer Ther. 2021 Jan-Dec;20:1534735420975853. doi: 10.1177/1534735420975853. PMID 33835869
- [Background] Jin Z, Lee C, Zhang K, Jeong R, Gan TJ, Richman DC. Utilization of Wearable Pedometer Devices in the Perioperative Period: A Qualitative Systematic Review. Anesth Analg. 2023 Apr 1;136(4):646-654. doi: 10.1213/ANE.0000000000006353. Epub 2023 Mar 16. PMID 36928149
- [Background] Wolk S, Linke S, Bogner A, Sturm D, Meissner T, Mussle B, Rahbari NN, Distler M, Weitz J, Welsch T. Use of Activity Tracking in Major Visceral Surgery-the Enhanced Perioperative Mobilization Trial: a Randomized Controlled Trial. J Gastrointest Surg. 2019 Jun;23(6):1218-1226. doi: 10.1007/s11605-018-3998-0. Epub 2018 Oct 8. PMID 30298422
- [Background] van Dijk-Huisman HC, Weemaes ATR, Boymans TAEJ, Lenssen AF, de Bie RA. Smartphone App with an Accelerometer Enhances Patients' Physical Activity Following Elective Orthopedic Surgery: A Pilot Study. Sensors (Basel). 2020 Aug 2;20(15):4317. doi: 10.3390/s20154317. PMID 32748876
- [Background] No JH, Kim K, Kim YB, Suh DH, Yang EJ, Hwang H, Yoo S. Effects of an activity tracker with feedback on physical activity in women after midline laparotomy: A randomized controlled trial. J Obstet Gynaecol Res. 2021 Jul;47(7):2544-2550. doi: 10.1111/jog.14807. Epub 2021 Apr 25. PMID 33899302